CLINICAL TRIAL: NCT04618913
Title: VICTORIE (VTE In Cancer - Treatment, Outcomes and Resource Use In Europe)
Brief Title: Anticoagulation in Patients With Venous Thromboembolism and Cancer
Acronym: VICTORIE
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661150; VICTORIE (Other: Alias Study Number)
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms; Embolism
Keywords: Venous thromboembolism; Eliquis; Neoplasms; Anti-Coagulation
MeSH Terms: conditions — Neoplasms; Embolism; Venous Thromboembolism | interventions — apixaban; Rivaroxaban; edoxaban; Dabigatran; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- VTE and history of cancer: VTE and history of cancer
  Interventions: Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban; Drug: Dabigatran; Drug: VKA; Drug: LMWH
- VTE and active cancer: VTE and active cancer
  Interventions: Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban; Drug: Dabigatran; Drug: VKA; Drug: LMWH

INTERVENTIONS:
Drug: Apixaban — Anticoagulant
Drug: Rivaroxaban — Anticoagulant
Drug: Edoxaban — Edoxaban
Drug: Dabigatran — Dabigatran
Drug: VKA — Vitamin K antagonist
Drug: LMWH — Low Molecular Weight Heparin

SUMMARY:
This study is a retrospective analysis of observational cohorts using data from prospectively collected administrative/claims data to investigate treatment patterns,healthcare resource utilisation (HCRU), direct and indirect costs (where feasible), and safety and effectiveness outcomes in patients with VTE and active cancer or patients with VTE and history of cancer who initiate anticoagulant treatment with a VKA, LMWH or NOACs.

ELIGIBILITY:
Inclusion Criteria:

* A VTE diagnosis
* Active cancer or history of cancer
* Treatment with VKA, NOAC (apixaban, rivaroxaban, dabigatran, edoxaban) or LMWH
* Age ≥ 18 years at the date of index VTE (Venous thromboembolic)

Exclusion Criteria:

* Prior VTE diagnosis
* Diagnosis of prior atrial fibrillation
* Inferior Vena Cava (IVC) filter
* Prior exposure to (OAC) oral anticoagulation or (PAC)parenteral anticoagulation - note: Prophylactic use of (OAC)/(PAC) allowed.
* Pregnancy
* More than one (OAC) oral anticoagulation or (PAC) parenteral anticoagulation dispensed on the index date.
* Patients with less than one day of follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of (VTE) venous thromboembolism and active cancer, or a history of cancer, being treated with anticoagulation.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Thromboembolism | 6 Months after treatment began as early as 1/1/2013
  The follow-up period during which outcome events of interest will be identified will run from the day after the index date until the end of the data collection or death, whichever occurs first. As data are updated at different times and frequencies in the different study countries, the date of the end of data collection will be determined after the relevant permissions have been acquired from the respective authorities.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661150